CLINICAL TRIAL: NCT03959306
Title: Effect of Black Seed Oil on Markers of Endothelial Dysfunction in Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy of Black Seed Oil in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amany Talaat Abdellatif El-Garf, Assistant Lecturer of Clinical Pharmacy, Faculty of Pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHCL14
Record Dates: First submitted 2019-05-18; First posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes Mellitus; Black Seed Oil; Endothelial Dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Nigella sativa oil; Hypoglycemic Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group I (Experimental): this group of patients will receive their standard anti-diabetic treatment in addition to 1800 mg of black seed oil soft gelatin capsule (900 mg twice daily) for three months
  Interventions: Dietary Supplement: Black Seed Oil; Drug: Anti-Diabetics
- Group II (Active Comparator): this group of patients will receive their standard anti-diabetic treatment only
  Interventions: Drug: Anti-Diabetics

INTERVENTIONS:
Dietary Supplement: Black Seed Oil — Black seed oil soft gelatin capsule
  Other Names: Nigella sativa oil
  Arms: Group I
Drug: Anti-Diabetics — standard anti-diabetic treatment prescribed for the patient

SUMMARY:
The purpose of this study is to determine the effect of black seed oil on markers of endothelial dysfunction in patients with type 2 diabetes mellitus .Also, to investigate its effect on glycemic control ,lipid profile and quality of life of those patients .

ELIGIBILITY:
Inclusion Criteria:

1. Age: adult patients with more than or equal 18 years old.
2. Previous diagnosis of Diabetes mellitus type 2 according to American Diabetes Association Criteria (ADA).
3. Approval to participate and give informed consent.

Exclusion Criteria:

1. Unstable coronary artery disease, cardiac arrhythmia or congestive heart failure.
2. Uncontrolled hypertension or recent stroke.
3. Chronic kidney disease or chronic liver disease.
4. Intake of black seed oil during the previous two months or any other antioxidant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-24 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Effect on Markers of Endothelial Dysfunction(The change in the level of soluble intercellular adhesion molecule ( ICAM) in serum using ELISA kit) | three months
  it will be assessed at baseline and after three months of treatment ( to determine the change from baseline at three months ) to determine whether it is effective in reducing marker of endothelial dysfunction (ICAM) in patients with type 2 diabetes mellitus

SECONDARY OUTCOMES:
Effect on Glycemic Control (Measurement of fasting blood glucose ) | three months
  it will be assessed at baseline and after three months of treatment to determine the anti-diabetic effect of black seed oil ( if it is effective in reducing fasting blood glucose from baseline)
Effect on Glycemic Control (Measurement of glycated hemoglobin) | three months
  it will be assessed at baseline and after three months of treatment to determine the anti-diabetic effect of black seed oil ( if it is effective in reducing glycated hemoglobin from baseline)
Effect on Lipid Profile ( Measurement of TC,TG, HDL-C,LDL-C) | three months
  it will be assessed at baseline and after three months of treatment
Effect on Inflammatory Status ( Measurement of High sensitive C-Reactive Protein using ELISA kit) | three months
  it will be assessed at baseline and after three months of treatment
Effect on Quality of Life ( Using Diabetes-39 questionnaire ) | three months
  it will be assessed at baseline and after three months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt